CLINICAL TRIAL: NCT01438541
Title: A Multi-centre, Post CE-mark, Open Study to Evaluate the Performance of Thin Self-adherent Dressing Coated With a Soft Silicone Layer on Subjects With High Risk of Category 2 or Above Pressure Ulceration
Brief Title: A Multi-centre Evaluation of the Performance of Window Dressings on Subjects With High Risk Pressure Ulceration
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Molnlycke Health Care AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Window 02
Record Dates: First submitted 2011-09-13; First posted 2011-09-22 (Estimated); Results first posted 2016-10-14 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2016-08

CONDITIONS: Pressure Ulcer
Keywords: No skin breakdown; Prevention; protection of the skin
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Window (Experimental): WindowTM is a protective layer that may reduce the shear and friction on the skin and may help to prevent skin breakdown. Window TM provides instant tack adhesion that minimizes the requirement of extra pressure in order to fixate well. The product does not leave residues and the adhesion level does not increase over time.
  Interventions: Device: Window

INTERVENTIONS:
Device: Window — Dressing

SUMMARY:
This study will be conducted in approximately 26 subjects in UK to yield 20 evaluable subjects at 3 sites with approximately 5-10 subjects/site. Subjects with acute vascular, surgical and orthopaedic medical care in the elderly admission, with a high risk to develop skin breakdown or subjects with category 1 pressure ulcer can be enrolled in this investigation.

The rational for this study is to evaluate the potential for Window in the prevention of pressure ulcers because of its ability to reduce shear and friction forces.

ELIGIBILITY:
Inclusion Criteria:

1. acute vascular, surgical, orthopaedic, medical or care of the elderly admission
2. aged 18 years or over
3. have an expected total length of stay of 5 or more days
4. at high risk of PU development due to one or more of the following

   * bedfast/chairfast AND completely immobile/very limited mobility
   * category 1 PU on any pressure area skin site (see appendix G)
5. give their written, informed consent to participate
6. expected to be able to comply with follow-up schedule

Exclusion Criteria:

1. risk area which doesn't fit the dressing size 6*7cm, 10*12 cm and 15*20cm
2. subject has category 2-4 pressure ulcer
3. subject has documented skin disease at time of enrolment, as judged by the investigator
4. known allergy/hypersensitivity to any of the components in the dressing
5. previous enroled in the present study
6. subject included in other ongoing clinical investigation at present, as judged by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2011-09; Primary Completion 2012-02 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carol Dealey, BSc, Principal Investigator — University Hospital Birmingham NHS
Locations (3):
- United Kingdom (3):
  - University Hospitals Birmingham NHS, Birmingham
  - Leeds General Infirmary, Leeds
  - The Mid Yourkshire Hospitals NHS Trust, Wakefield

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period was from 03 October 2011-21 February 2012. The study was conducted at three wound care units in United Kingdom.
Pre-assignment Details: There was no wash-out or run-in phase included in the study.
Groups:
- Window: WindowTM is a protective layer that may reduce the shear and friction on the skin and may help to prevent skin breakdown.
Period: Overall Study
Arm/Group | Window
Started | 29
Completed | 22
Not Completed | 7
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 1
Not completed — discharge from the hospital | 5

BASELINE CHARACTERISTICS:
Arm/Group | Window
Number analyzed (Participants) | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.6 (16.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 9
Region of Enrollment [Number; unit: participants]
  United Kingdom | 29

OUTCOME MEASURES:

1. Primary Outcome: Erythema ( No/Yes)
Description: Total improvement of erythema
Time Frame: 14 days
Population: Vulnerable subjects with high risk of skin breakdown.
Measure: Number; unit: participants
Arm/Group | Window
Number analyzed (Participants) | 29
participants
  Erytehma Baseline No | 5
  Erytema Baseline Yes | 24
  Erythema Last visit No | 16
  Erytehma Last visit Yes | 13

2. Secondary Outcome: Overall Experience of Use of the Dressing
Description: Investigator and Nurses evaluate the overall Experience of using of the dressing rated on a scale from Very Poor, Poor,Good, Very Good, Excellent, Not measured
Time Frame: 14 days
Measure: Number; unit: participants
Arm/Group | Window
Number analyzed (Participants) | 29
participants
  Very Poor | 1
  Poor | 10
  Good | 15
  Very Good | 0
  Excellent | 1
  Not measured | 2

3. Secondary Outcome: Evaluate the Dressing Shape
Description: Investigator and Nurses evaluated the shape of the dressing rated on a scale from Very Poor, Poor,Good, Very Good, Excellent
Time Frame: 14 days
Measure: Number; unit: participants
Arm/Group | Window
Number analyzed (Participants) | 29
participants
  Very Poor | 0
  Poor | 4
  Good | 22
  Very Good | 1
  Excellent | 2

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from baseline to termination (14days)
Arm/Group | Window
Serious Adverse Events (participants affected / at risk) | 0/29
Other Adverse Events (participants affected / at risk) | 2/29
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Window (N=29)
Ruptured blister - broken skin (Skin and subcutaneous tissue disorders) | 1 (1)
Recurrence of ruptured blister in different (Skin and subcutaneous tissue disorders) | 1 (1)
Grade 2 area to L buttock 2mm x 2 mm (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No